CLINICAL TRIAL: NCT02174263
Title: Tocilizumab in Chronic GVHD Refractory to at Least Two Prior Therapies
Brief Title: Tocilizumab for Chronic Graft-versus-Host Disease Treatment
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study never opened due to lack of funds.
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 9130; NCI-2014-01204 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9130 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2014-06-23; First posted 2014-06-25 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Graft Versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — tocilizumab; Immunoglobulin G; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (tocilizumab) (Experimental): Patients receive tocilizumab IV over 1 hour every 2 weeks for 12 weeks (weeks 1, 3, 5, 7, 9, and 11) and then every 4 weeks for 12 weeks (weeks 13, 17, and 21).
  Interventions: Biological: tocilizumab; Other: laboratory biomarker analysis; Other: quality-of-life assessment

INTERVENTIONS:
Biological: tocilizumab — Given IV
  Other Names: Actemra; immunoglobulin G1, anti-(human interleukin 6 receptor) (human-mouse monoclonal MRA heavy chain), disulfide with human-mouse monoclonal MRA kappa chain dimer; MRA; R-1569; RoActemra
Other: laboratory biomarker analysis — Correlative studies
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This phase II trial studies how well tocilizumab works in treating chronic graft-versus-host disease (GVHD) in patients that have not responded to treatment after at least two prior therapies. Tocilizumab blocks a protein that stimulates the body's immune system. By blocking this protein, the investigators may reduce the symptoms of chronic GVHD.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Efficacy will be determined by the proportion of patients with failure free survival (FFS) at 6 months.

SECONDARY OBJECTIVES:

I. Patients achieving a complete response (CR) or partial response (PR) at 6 months based on clinician judged response.

II. Patients achieving a CR or PR by objective response measures at 6 months.

III. Failure-free survival (FFS) at 1 year.

IV. Change in steroid dose from enrollment to 6 months (mo).

TERTIARY OBJECTIVES:

I. Biologic studies will be done to determine possible mechanisms of response.

OUTLINE:

Patients receive tocilizumab intravenously (IV) over 1 hour every 2 weeks for 12 weeks (weeks 1, 3, 5, 7, 9, and 11) and then every 4 weeks for 12 weeks (weeks 13, 17, and 21).

After completion of study treatment, patients are followed up at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject has moderate or severe overlap chronic (c)GVHD according to National Institutes of Health (NIH) criteria
* Active cGVHD despite treatment with at least two immunosuppressive treatments (not including GVHD prophylaxis) in the past year
* Subject underwent allogeneic stem cell transplantation at least 6 months prior to enrollment
* Subject has not started any new systemic immunosuppressive therapies within 2 weeks prior to enrollment
* Female subjects of child bearing potential must have a negative pregnancy test prior to first dose of tocilizumab and must agree to practice effective contraception during the study
* Subject meets the following medication restriction requirements and agrees to follow medication restrictions during the study; the following concomitant medications are not allowed: cyclophosphamide, abatacept, etanercept, adalimumab infliximab, golimumab, tofacitinib, and alemtuzumab; these medications also cannot have been used for 5 half-lives prior to enrollment
* Subject agrees to comply with the study requirements and agrees to come to the clinic for required study visits

Exclusion Criteria:

* Donor lymphocyte infusion in the preceding 100 days
* Subject has bronchiolitis obliterans, bronchiolitis obliterans with organizing pneumonia or cryptogenic organizing pneumonia as the sole manifestation of cGVHD
* Uncontrolled bacterial, viral infection or invasive fungal infection
* Evidence of malignancy within 6 months of study enrollment; this is defined as clear morphologic, radiologic or molecular evidence of disease; mixed chimerism is allowed at the discretion of the clinician
* Treatment with any non-Food and Drug Administration (FDA) approved agent within 4 weeks (or 5 half-lives of the investigational drug, whichever is longer) of study enrollment
* Immunization with a live, attenuated vaccine within 4 weeks prior to study enrollment
* History of severe allergic or anaphylactic reactions to human, humanized or murine monoclonal antibodies
* Tuberculosis requiring treatment within the past 3 years; all patients must have a negative quantiferon test within 4 weeks prior to starting study drug
* Pregnant or breast-feeding women
* Patients (both men and women) with reproductive potential not willing to use an effective method of contraception
* Serum creatinine > 1.6 mg/dL (141 umol/L) in females and > 1.9 mg/dL (168 umol/L) in males; patients with serum creatinine values exceeding these limits are eligible for the study if their estimated glomerular filtration rates (GFR) are > 30 ml/min/1.73 m^2
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 1.5 times upper limit of normal (ULN)
* Total bilirubin > upper limit of normal (ULN)
* Absolute neutrophil count < 1.5 x 10^9/L (1500/mm^3)
* Known active hepatitis B or C; patients must have a negative test for hepatitis B surface antigen, hepatitis B core antibody and hepatitis C antibody within 4 weeks prior to starting study drug
* Known uncontrolled cytomegalovirus (CMV) polymerase chain reaction (PCR) reactivation per institutional standards; once CMV has been treated and stable per institutional standards, patient may be enrolled; CMV PCR will be tested within two weeks prior to starting study drug
* History of diverticulitis, Crohn's disease or ulcerative colitis
* History of demyelinating disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
FFS | At 6 months

SECONDARY OUTCOMES:
Patients achieving CR or PR based on objective measures, as recommended by the NIH Consensus Conference for chronic GVHD | At 6 months
Patients achieving a CR or PR based on clinician judged response | At 6 months
Relative change in daily prednisone dose | Baseline to 6 months
  Prednisone is not a pre-specified intervention; however, some patients may take prednisone while on this study.

OTHER OUTCOMES:
B cell subsets | Up to week 21
Tumor necrosis factor (ligand) superfamily, member 13b (BAFF) levels | Up to week 21
T cell subsets | Up to week 21

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Lee, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (5):
- United States (5):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic, Rochester, Minnesota
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin